CLINICAL TRIAL: NCT04053101
Title: Role of FDG-PET CT in the Management of Muscle Invasive Bladder Cancer
Acronym: TEP-Vessie
Status: Completed | Type: Observational
Sponsor: Institut Bergonié (Other)
Responsible Party: Sponsor
Other Study IDs: IB2018-TEP vessie; MR 3316040319 (Other: Institut National des Données de Santé (INDS))
Record Dates: First submitted 2019-07-04; First posted 2019-08-12 (Actual); Results first posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Muscle Invasive Bladder Cancer
Keywords: Bladder cancer; PET CT; CT scan; Lymph node staging; TNM staging
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MIBC: Patients with muscle invasive bladder cancer (MIBC)
  Interventions: Device: PET CT

INTERVENTIONS:
Device: PET CT — Every patient undergoing a PET CT at the time of diagnosis of muscle invasive bladder cancer from January 2005 to December 2017 in Bordeaux (Institut Bergonié and University Hospital).

SUMMARY:
Bladder cancer is the seventh cause of cancer mortality in France. Overall survival is poor, between 45 and 50% at 5 years.

Optimal staging of lymph nodes and metastasis is crucial for treatment decision of muscle invasive bladder cancer (MIBC).

Guidelines do not recommend FDG-Positron Emission Tomography (PET) Computed Tomography (CT), but rather CT for lymph node and metastatic staging, despite its low accuracy. We performed a retrospective analysis of patients undergoing PET CT for localized MIBC in two centers, to help define the utility of PET CT in this setting.

DETAILED DESCRIPTION:
Background:

Bladder cancer is the second most frequent genito-urinary cancer, and the seventh cause of cancer mortality in France. Overall survival is poor, between 45 and 50% at 5 years. Curative treatment of muscle invasive urothelial carcinoma localized to the bladder includes cisplatin-based neoadjuvant chemotherapy, followed by radical cystectomy with lymph nodes dissection. Nonetheless, surgery indications depend on pre-operative staging regarding nodes and metastatic involvement.

Computed Tomography (CT) scan is the reference imaging study for loco-regional and metastatic staging. Lymph node involvement evaluation is based on morphologic criteria only. Its sensitivity lies between 30 and 53% and its specificity between 67 and 91%. Yet, optimal node staging is crucial for therapeutic decision.

FDG-Positron Emission Tomography (PET) CT, using both morphologic and functional criteria, could help for node staging in muscle invasive bladder cancer assessment, especially by detecting infracentimetric involved lymph nodes. Moreover, it could be useful for detecting distant metastasis.

Objective: To evaluate the accuracy of the PET CT for lymph node staging and to determine the rate of treatment modification according to PET CT results Methods: Retrospective study based on the medical records of every patient undergoing a PET CT at the time of diagnosis of MIBC from 01/2005 to 12/2017 in Bordeaux (Bergonie Institute and University Hospital). PET CT could have been done before any treatment (PET 1) and/or after neo-adjuvant chemotherapy and before surgery (PET 2).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Muscle Invasive Urothelial Carcinoma of the bladder (classified at least pT2 on TURB)
* Diagnosis between January 2005 and December 2017
* PET CT done during initial assessment before surgery (at the time of diagnosis and/or after neoadjuvant chemotherapy)
* Management of cancer at Institut Bergonié or at Bordeaux University Hospital
* Previous treatment for Non Muscle Invasive Bladder Cancer allowed

Exclusion Criteria:

* Management of cancer outside of Institut Bergonié or Bordeaux University Hospital
* No PET CT done during initial assessment (before surgery)
* Rare pathological type of bladder cancer without urothelial carcinoma (epidermoid carcinoma, neuro-endocrine carcinoma, …)
* Extra-vesical urothelial carcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Every patient undergoing a PET CT at the time of diagnosis of muscle invasive bladder cancer from January 2005 to December 2017 in Bordeaux (Institut Bergonié and University Hospital).
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre Hospitalier Universitaire de Bordeaux, Bordeaux
  - Institut Bergonie, Bordeaux

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bertolaso P, Brouste V, Cazeau AL, de Clermont-Gallerande H, Bladou F, Cabart M, Lefort F, Gross-Goupil M. Impact of 18 FDG- PET CT in the Management of Muscle Invasive Bladder Cancer. Clin Genitourin Cancer. 2022 Jun;20(3):297-297.e6. doi: 10.1016/j.clgc.2022.01.009. Epub 2022 Jan 14. PMID 35101381

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MIBC
Started | 130
Completed | 130
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | MIBC
Number analyzed (Participants) | 130
Age, Continuous [Median (Full Range); unit: years] | 66 [43 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 113
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 130

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of the PET CT for Lymph Node Staging in Terms of Sensitivy Rate
Description: Performance sensitivity of FDG-PET CT for LN staging on diagnosis of MIBC (before and after NAC and before cystectomy and LN dissection).
  Gold standard : pathological results (complete response vs no complete response).
  Comparison of PET-CT TNM staging between patients with and patients without a Pathological Complete Response.
  Sensitivity rate : count of participants with complete response as per FDG-PET divided by count of participants with pathoplogical complete response
Time Frame: 16 weeks after inclusion
Population: Patients with complete pathological response
Measure: Count of Participants; unit: Participants
Groups:
- Eligible MIBC Patients: Patients with pelvic LN dissection and with a FDG-PET CT before neoadjuvant chemotherapy
Arm/Group | Eligible MIBC Patients
Number analyzed (Participants) | 26
Participants | 21

2. Primary Outcome: Accuracy of the PET CT for Lymph Node Staging in Terms of Specificity Rate
Description: Performance specificity of FDG-PET CT for LN staging on diagnosis of MIBC (before and after NAC and before cystectomy and LN dissection).
  Gold standard : pathological results (complete response vs no complete response).
  Comparison of PET-CT TNM staging between patients with and patients without a Pathological Complete Response Specificiity rate : count of participants with NO complete response as per FDG-PET divided by count of participants with NO pathoplogical complete response
Time Frame: Date of pathological results, up to 20 weeks after inclusion
Population: Participants with NO pathoplogical complete response
Measure: Number; unit: participants
Arm/Group | Eligible MIBC Patients
Number analyzed (Participants) | 59
participants | 32

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious Adverse Events and Other (Not Including Serious) Adverse Events were not collected
Description: All-Cause Mortality, Serious Adverse Events and Other (Not Including Serious) Adverse Events were not collected
Arm/Group | MIBC
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-05): https://cdn.clinicaltrials.gov/large-docs/01/NCT04053101/Prot_SAP_000.pdf